CLINICAL TRIAL: NCT06395558
Title: Internet-Based Interventions for Cardiac Arrest Survivors
Acronym: ENFORCER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ENFORCER
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairment; Depression, Anxiety; Cardiac Arrest; Quality of Life; Social Functioning; Sexual Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Anxiety Disorders; Heart Arrest; Social Adjustment; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be unaware about the study arm allocation of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention (Experimental)
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle intervention — Multimodal web-based intervention programme on anxiety, depression and cognitive impairment consisting of knowledge development sessions and practical/gaming sessions focused on different domains: cognitive competence, socio-relational competence and emotions/affectivity, and physical activity-nutrition
  Arms: Lifestyle intervention

SUMMARY:
Anxiety, depression and cognitive impairment symptoms are common among cardiac arrest survivors. This randomized clinical trial will test whether an internet-based lifestyle intervention administered through a web app can foster anxiety and depression symptoms in patients who survived an out-of-hospital cardiac arrest and suffer from these symptoms

ELIGIBILITY:
Inclusion Criteria:

* Hospital discharge after out-of-hospital cardiac arrest with Cerebral Performance Category 1 or 2
* HADS anxiety or depression ≥ 8 and/or TICS ≤ 31
* Informed consent for participation in the study
* Native Italian speaker or adequate understanding of the Italian language
* Adequate ability to use the web to guarantee access to the contents

Exclusion Criteria:

* Previous cognitive dysfunction
* Previous psychiatric disease
* Previous episode of out-of-hospital cardiac arrest

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 12 months
  HADS (Hospital Anxiety and Depression Scale) score < 8 for depression or anxiety and TICS (Telephone Interview for Cognitive Status) > 31

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) value | 12 months
  Depression and anxiety symptoms
TICS (Telephone Interview for Cognitive Status) | 12 months
  Cognitive symptoms
SF-12 (Short Form Health Survey 36) | 12 months
  Health Related Quality of Life
NRS (Neurobehavioural rating scale), PCRS (Patient Competency Rating Scale) | 12 months
  Behavioural symptoms
NRS (Neurobehavioural rating scale) | 12 months
  Behavioural symptoms
Pittsburgh Sleep Quality Index (PSQI) | 12 months
  Sleep Quality
Sexual Interest and Satisfaction Scale (SISS) | 12 months
  Sexual Interest and Satisfaction
Zarit Burden Inventory (ZBI) | 12 months
  Caregiver Burden
PCRS (Patient Competency Rating Scale) | 12 months
  Behavioural symptoms
HADS (Hospital Anxiety and Depression Scale) - Caregiver | 12 months
  Caregiver's depression and anxiety symptoms
PSQI (Pittsburgh Sleep Quality Index) - Caregiver | 12 months
  Caregiver's sleep quality
SF-12 (Short Form Health Survey 36) - Caregiver | 12 months
  Caregiver's Health Related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gamberini, MD, Principal Investigator — Azienda USL Bologna
Locations (2):
- Italy (2):
  - Montecatone Rehabilitation Institute, Imola, Bologna
  - Azienda Unità Sanitaria Locale, Bologna

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized patient data will be shared in an online repository
Supporting Information: Study Protocol
Time Frame: After study publication, indefinitely.
Access Criteria: No Access restrictions

REFERENCES:
- [Derived] Gamberini L, Rucci P, Dolcini C, Masi M, Simoncini L, Tartaglione M, Del Giudice D, Domina R, Fagiolini A, Salucci P; Collaborators. ENFORCER, internet-based interventions for cardiac arrest survivors: A study protocol for a randomised, parallel-group, multicentre clinical trial. Resusc Plus. 2024 Sep 18;20:100772. doi: 10.1016/j.resplu.2024.100772. eCollection 2024 Dec. PMID 39328897